CLINICAL TRIAL: NCT00401232
Title: Blood Collection In Healthy Adult Volunteers To Obtain Serum For Use In Serum Bactericidal Activity Assay Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 6108A1-800; B1971032 (Other: Alias Study Number)
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Blood Collection

INTERVENTIONS:
Procedure: Blood Collection — Blood Collection

SUMMARY:
This is a study to collect blood from volunteers to assist in assay development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers aged 18-64

Exclusion Criteria:

* Bleeding disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 955 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
"No outcome measures". Blood collected for assay development. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - SNBL Clinical Pharmacology Center, Baltimore, Maryland
  - Frontage Clinical Services Inc, Hackensack, New Jersey

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6108A1-800&StudyName=Blood%20Collection%20In%20Healthy%20Adult%20Volunteers%20To%20Obtain%20Serum%20For%20Use%20In%20Serum%20Bactericidal%20Activity%20Assay%20Development